CLINICAL TRIAL: NCT03482271
Title: Analysing Emergency and Urgent Care System Demand in Yorkshire and Humber: A Data-linkage Study of Pre-hospital, Emergency Department and Out of Hours Service Data
Brief Title: Connected Yorkshire: A Data-linkage Study of Pre-hospital, Emergency Department and Out of Hours Service Data
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sheffield (Other)
Collaborators: Northern Health Science Alliance (NHSA) (Unknown)
Responsible Party: Principal Investigator, Professor Suzanne Mason, Proessor of Emergency Medicine, University of Sheffield
Other Study IDs: USheffield
Record Dates: First submitted 2018-03-15; First posted 2018-03-29 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Emergency and Urgent Care Pathways
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention - data collection only — No intervention - data collection only

SUMMARY:
There is increased demand on emergency departments (ED) across the UK. The services are becoming stretched and as a result waiting times are increasing and patient care is suffering.

By linking together patient data from different hospitals and services across Yorkshire, researchers are able to build a more complete picture of how emergency and urgent care (UEC) services in the region function.

This picture will help researchers understand the flow of patients through EUC services, to understand what the most common health issues are and to better plan community services in the future. The anonymous data can help scientists understand EUC services across an entire region and suggest improvements in a much more synchronised way.

Health service managers will also be able to understand how one ED in Yorkshire compares to another. By re-using existing data researchers will also allow hospitals to learn lessons from each other so that each local service can improve and deliver better care for its patients.

In the future, this information will help researchers to plan ahead and forecast disease outbreaks. The data used will, over time, tell a story that will help deliver better and more targeted care.

The aim of the research project is to build a unique dataset based on expertise already being developed across the Yorkshire and Humber region. We will collect routine NHS data from a number of providers of EUC and link the data to provide a coherent picture of EUC demand. This rich data source will allow the EUC services to be viewed as a whole system, enabling demand on the system by patients to be analysed as well as the flow of patients through the system.

ELIGIBILITY:
Inclusion Criteria:

* access urgent and emergency care services in Yorkshire and the Humber region between 2011 and 2017

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Any person who has accessed an urgent and emergency care service in Yorkshire and the Humber region between 2011 and 2017
Sampling Method: Non-Probability Sample
Enrollment: 7500000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
NHS111 | 2011-2017
  Number of people accessing NHS111 and transferred to the emergency department by the Yorkshire Ambulance Service, stratisfied by age, gender, presenting complaint, location

SECONDARY OUTCOMES:
YAS | 2011-2017
  Number of people accessing the Yorkshire Ambulance Service and transferred to the emergency department, stratisfied by age, gender, presenting complaint, location
Direct ED | 2011-2017
  Number of people accessing the emergency department (directly), stratisfied by age, gender, presenting complaint, location

OTHER OUTCOMES:
Mapping of UEC service use | 2011-2017
  Using the linked data, map how the UEC service is used by patients. How far people will travel to attend the ED; Where are people travelling from (home, etc), the flow through each of the services throughout the time period covered (annually, monthly, daily, hourly), etc

IPD SHARING:
Plan to Share IPD: Yes
The study is now a Research Database and researchers can obtain data extracts, on application, for use in research aligned with the CHC study focus.
Supporting Information: Study Protocol
Time Frame: 2019
Access Criteria: Contact Maxine Kuczawski for details
URL: https://www.sheffield.ac.uk/scharr/sections/hsr/cure/chc/study